CLINICAL TRIAL: NCT05554354
Title: Phase 2 Trial of Fulvestrant and Binimetinib in Patients With Hormone Receptor-Positive Metastatic Breast Cancer With Inactivating or Inferred Inactivating NF1 Alterations: A ComboMATCH Treatment Trial
Brief Title: Testing the Use of Fulvestrant and Binimetinib Targeted Treatment for NF1 Mutation in Hormone Receptor-Positive Metastatic Breast Cancer (A ComboMATCH Treatment Trial)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Other - slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-07265; NCI-2022-07265 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY191-N2 (Other: NRG Oncology); EAY191-N2 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-09-22; First posted 2022-09-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic HER2-Negative Breast Carcinoma; Metastatic Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: interventions — binimetinib; Biopsy; Specimen Handling; Fulvestrant; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort I (Arm I) (fulvestrant, binimetinib) (Experimental): Patients receive fulvestrant IM on day 1 and day 15 of cycle 1 and day 1 of subsequent cycles and binimetinib PO BID on days 15 to 28 of cycle 1 and day 1 through 28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a CT, MRI, or bone scan, ECHO or MUGA, and tumor biopsy, as well as possible blood sample collection during screening and on study.
  Interventions: Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan
- Cohort I (Arm II) (Active Comparator): Patients receive fulvestrant IM on day 1 and day 15 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who progress on fulvestrant alone may migrate to cohort II if they meet the migration eligibility criteria. Patients not willing to migrate to cohort II will have further therapy at the investigator's discretion. Patients undergo a CT, MRI, or bone scan and tumor biopsy, as well as ECHO or MUGA and possible blood sample collection during screening and on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan
- Cohort II (fulvestrant, binimetinib) (Experimental): Patients receive fulvestrant IM on day 1 of each cycle and binimetinib PO BID on days 15-28 of cycle 1 and day 1 through 28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT, MRI, or bone scan, ECHO or MUGA and tumor biopsy, as well as possible blood sample collection during screening and on study.
  Interventions: Drug: Binimetinib; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Fulvestrant; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Drug: Binimetinib — Given PO
  Other Names: ARRY 162; ARRY 438162; ARRY-162; ARRY-438162; ARRY162; ARRY438162; MEK 162; MEK-162; MEK162; Mektovi
  Arms: Cohort I (Arm I) (fulvestrant, binimetinib); Cohort II (fulvestrant, binimetinib)
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fulvestrant — Given IM
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ICI-182780; ICI182780; ZD 9238; ZD-9238; ZD9238
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning

SUMMARY:
This phase II ComboMATCH treatment trial compares the usual treatment alone (fulvestrant) to using binimetinib plus the usual treatment in patients with hormone receptor positive breast cancer that has spread from where it first started to other places in the body (metastatic) and has an NF1 genetic change. Fulvestrant is a hormonal therapy that binds to estrogen receptors in tumor cells, resulting in estrogen receptor destruction and decreased estrogen binding, which may inhibit the growth of estrogen-sensitive tumor cells. Binimetinib is a targeted therapy that may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. The addition of binimetinib to fulvestrant in breast cancers with an NF1 genetic change could increase the percentage of tumors that shrink as well as lengthen the time that the tumors remain stable (without progression) as compared to fulvestrant alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether the combination of fulvestrant and binimetinib improves progression-free survival (PFS) compared to treatment with fulvestrant alone in patients not previously treated with fulvestrant. (Cohort 1) II. To determine whether overall response rate (ORR) within 4 months in patients who have previously progressed on a fulvestrant-containing regimen is greater than 10%, as a historical comparison, when these patients receive combination fulvestrant and binimetinib therapy. (Cohort 2)

SECONDARY OBJECTIVES:

I. To estimate ORR at any time after the start of the treatment for Cohort 2 and separately for the two arms in Cohort 1.

II. To estimate PFS distribution in Cohort 2. III. To estimate clinical benefit rate separately for the two arms in Cohort 1 and Cohort 2.

IV. To determine the safety and toxicity profile in both cohorts. V. To estimate the overall survival (OS) in both cohorts. VI. Collect tissue and provide it to the ComboMATCH Registration Protocol to assess concordance between the diagnostic tumor mutation profile generated by the Designated Laboratories, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor deoxyribonucleic acid (DNA) (ctDNA) mutation profile from plasma, as described in ComboMATCH Registration Protocol. For this treatment substudy, the outcome objective will be to report the proportion of cases providing sufficient tissue for that integrated scientific activity in the ComboMATCH Registration Protocol.

EXPLORATORY BIOMARKER OBJECTIVES:

I. To analyze the cell-free (cf)DNA at progression to determine the changes in cfDNA profile in order to understand blood-based mutation dynamics.

II. To analyze RNAseq at progression to determine potential pathways that are altered that may contribute to the sensitivity/resistance.

III. To discover/detect novel biomarkers using microscaled proteogenomics by analyzing the proteins and phosphor-proteins along with genomics to determine potential pathways that may correlate with the response to the combination treatment.

IV. To detect the loss of NF1, using immunohistochemistry staining to precisely measure the level of the NF1 protein.

V. To determine the variant allele frequency (VAF) of mutant NF1 measuring by using droplet digital polymerase chain reaction (ddPCR) for the targeted NF1 gene level.

OUTLINE: Patients who are fulvestrant naive are assigned to Cohort I, while patients who are fulvestrant resistant are assigned to Cohort II.

COHORT I: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive fulvestrant intramuscularly (IM) on day 1 and day 15 of cycle 1 and day 1 of subsequent cycles and binimetinib orally (PO) twice daily (BID) on days 15 to 28 of cycle 1 and day 1 through 28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo a computed tomography (CT), magnetic resonance imaging (MRI), or bone scan, echocardiography (ECHO) or multi-gated acqusition scan (MUGA), and tumor biopsy, as well as possible blood sample collection during screening and on study.

ARM II: Patients receive fulvestrant IM on day 1 and day 15 of cycle 1 and day 1 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who progress on fulvestrant alone may migrate to cohort II if they meet the migration eligibility criteria. Patients not willing to migrate to cohort II will have further therapy at the investigator's discretion. Patients undergo a CT, MRI, or bone scan and tumor biopsy, as well as ECHO or MUGA and possible blood sample collection during screening and on study.

COHORT II: Patients receive fulvestrant IM on day 1 of each cycle and binimetinib PO BID on days 15-28 of cycle 1 and day 1 through 28 of subsequent cycles. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo a CT, MRI, or bone scan, ECHO or MUGA and tumor biopsy, as well as possible blood sample collection during screening and on study.

Upon completion of study treatment patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have enrolled onto EAY191 and must have been given a treatment assignment to ComboMATCH to EAY191-N2 based on the presence of an actionable mutation as defined in EAY191
* The patient must be enrolled on the ComboMATCH Master Registration Trial EAY191

  * Note: Patients must fulfill all eligibility criteria outlined in the ComboMATCH Registration Trial EAY191 at the time of registration to EAY191-N2. This includes submission of next-generation sequencing (NGS) data from one of the National Cancer Institute (NCI) credentialed designated laboratories for all potential patients prior to treatment trial assignment. Copy number and allele frequency cutoff as per the Registration protocol
* Patients must have disease that can be safely biopsied and agree to a pre-treatment biopsy or, if disease cannot be safely biopsied, have archival tissue available from within 12 months prior to the date of registration on the ComboMATCH registration trial (EAY191)

  * Please note the current actionable marker of interest (aMOI)/actionable alteration list for this treatment trial can be found on the Cancer Trial Support Unit (CTSU) ComboMATCH Registration protocol page
  * Please note novel/Dynamic aMOI can be submitted for review per the process described in the ComboMATCH Registration protocol
* A COMBOMATCH TREATMENT TRIAL EAY191-N2 ELIGIBILITY CRITERIA:
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Histologically or cytologically confirmed invasive breast carcinoma
* Confirmed metastatic disease by either imaging or tissue diagnosis
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and one additional lesion that can be biopsied (primary, metastatic both allowed)
* Patients must have inactivating or inferred inactivating NF1 alterations detected in tumor as determined by the ComboMATCH screening assessment
* The tumor must have been determined to be estrogen receptor (ER) and/or progesterone receptor (PgR) positive assessed by current American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guideline recommendations for hormone receptor testing. Patients with >= 1% ER or PgR staining by immunohistochemistry (IHC) are considered positive
* The tumor must have been determined to be HER2-negative by current ASCO/CAP guidelines
* Prior use of CDK4/6 inhibitor(i) is required
* Prior use of fulvestrant regardless of duration is allowed and will determine treatment assignment
* Up to one line of chemotherapy in metastatic setting is allowed
* Absolute neutrophil count >= 1,500/mm^3
* Platelet count >= 100,000/ mm^3
* Hemoglobin level >= 10 g/dL
* Creatinine clearance (CrCL) of ≥ 30 mL/min by the Cockcroft-Gault formula
* Total bilirubin level =< institutional upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) must be =< 5.0 x ULN
* For patients who will be assigned to Cohort 2 (fulvestrant-resistant), a left ventricular ejection fraction (LVEF) assessment must be performed within 12 weeks prior to registration. The LVEF must be >= 50% regardless of the cardiac imaging facility's lower limit of normal. (LVEF assessment performed by echocardiogram is preferred; however, MUGA scan may be substituted based on institutional/situational preferences)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial
* ELIGIBILITY CRITERIA FOR COHORT 1, TREATMENT REGIMEN 2 PATIENTS WHO MIGRATE TO COHORT 2: Cohort migration: Patients treated with control treatment fulvestrant who experience disease progression may be eligible to migrate to Cohort 2 and receive combination treatment with binimetinib and fulvestrant. Patients who choose to do so must meet laboratory values and performance status requirements below and should begin treatment within 28 days
* PATIENTS WHO MIGRATE TO COHORT 2: Patient's willingness to migrate to Cohort 2 affirmed
* PATIENTS WHO MIGRATE TO COHORT 2: The patient must have an ECOG performance status of 0-2
* PATIENTS WHO MIGRATE TO COHORT 2: Absolute neutrophil count >= 1,500/mm^3
* PATIENTS WHO MIGRATE TO COHORT 2: Platelet count >= 100,000/ mm^3
* PATIENTS WHO MIGRATE TO COHORT 2: Hemoglobin level >= 10 g/dL
* PATIENTS WHO MIGRATE TO COHORT 2: Total bilirubin level =< institutional upper limit of normal (ULN)
* PATIENTS WHO MIGRATE TO COHORT 2: AST and ALT must be =< 5.0 x ULN
* PATIENTS WHO MIGRATE TO COHORT 2: Creatinine clearance (CrCL) of ≥30 mL/min by the Cockcroft-Gault formula
* PATIENTS WHO MIGRATE TO COHORT 2: A LVEF performed within the last 3 months must be >= 50% regardless of the cardiac imaging facility's lower limit of normal (LVEF assessment performed by echocardiogram is preferred; however, MUGA scan may be substituted based on institutional/situational preferences)
* PATIENTS WHO MIGRATE TO COHORT 2: Pregnancy test according to institutional standards must be negative (for patients of childbearing potential only)

Exclusion Criteria:

* Concurrent anticancer therapy
* Active autoimmune disease requiring systemic treatment within the past 3 months, documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents
* Active brain metastasis. Brain metastases that have been stable for at least 1 month after completion of treatment are not an exclusion criterion
* History of or evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment/central serous, chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration
* Patients will be excluded if they currently have the following risk factors for RVO that are documented prior to the enrollment:

  * Known uncontrolled glaucoma with intra-ocular pressures >= 21 mmHg
  * Known serum cholesterol >= grade 2.
  * Known hypertriglyceridemia >= grade 2
  * Known hyperglycemia (fasting) >= grade 2
* Patients with baseline QT corrected for heart rate (QTc) > 500 ms, either induced by medication or congenital long QT syndrome will be excluded due to known side effects of binimetinib
* Nervous system disorder (paresthesia, peripheral motor neuropathy, or peripheral sensory neuropathy) >= grade 2
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements or interfere with interpretation of study results
* Pregnancy or lactation at the time of registration or intention to become pregnant during the study (Note: Pregnancy testing according to institutional standards for patients of childbearing potential)

  * For binimetinib, highly effective contraception should be used for at least 30 days after the last dose, and patients should not breastfeed for 3 days after the last dose
  * For fulvestrant, highly effective contraception should be used for 1 year after the last dose, and patients should not breastfeed for 1 year after the last dose
* Use of any investigational product within 30 days prior to study entry
* INELIGIBILITY CRITERIA FOR COHORT 1, TREATMENT REGIMEN 2 PATIENTS WHO MIGRATE TO COHORT 2
* PATIENTS WHO MIGRATE TO COHORT 2: Not a candidate for binimetinib in the opinion of the treating investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-09-13 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) (Cohort I) | The duration between randomization and progression or death from all cause, whichever happens first, assessed up to 5 years
  PFS of the two study arms will be compared by log-rank test (1-sided, alpha=0.1). Kaplan-Meier plot will be provided. Hazard ratio (HR) and the corresponding 95% confidence interval (CI) will be estimated by Cox proportional model using treatment as covariate.
Objective response rate (ORR) (Cohort II) | Within 4 months of the start of treatment
  ORR is the percentage of patients who reaches a complete or partial response (defined by Response Evaluation Criteria in Solid Tumors [RECIST] version[v]1.1) within 4 months of the start of the treatment. ORR will be calculated as the proportion of patients achieved partial response (PR) or complete response (CR) within 4 months after the initiation of the treatment. ORR will be reported with corresponding 95% exact CI. Patients who have withdrawn from the study before any efficacy follow up are considered non-evaluable for clinical response and will be replaced.

SECONDARY OUTCOMES:
ORR for each study arm (Cohort I) | Any time after the start of the treatment, assessed up to 5 years
  ORR is the percentage of patients who reach a complete or partial response (defined by RECIST v1.1) any time after the start of the treatment. ORR for each study arm will be calculated with corresponding 95% exact CI. Fisher exact test will be used to compare the ORR of the two study arms.
ORR (Cohort II) | Any time after the start of the treatment, assessed up to 5 years
  ORR is the percentage of patients who reach a complete or partial response (defined by RECIST v1.1) any time after the start of the treatment.
Clinical benefit rate | Any time after the start of the treatment, assessed up to 5 years
  Defined as proportion of patients who achieved a CR, PR, or stable disease defined by RECIST criteria any time after the start of the treatment. Clinical benefit rate will be analyzed for each arm of cohort I and cohort II as described for ORR. ORR for each study arm will be calculated with corresponding 95% exact CI. Fisher exact test will be used to compare the ORR of the two study arms.
PFS (Cohort II) | The duration between randomization and progression or death from all cause, whichever happens first, assessed up to 5 years
  PFS for cohort II will be summarized using the Kaplan-Meier's method. Median PFS with corresponding 95% CI will be provided.
Overall survival (OS) | The duration between randomization and death of all causes, assessed up to 5 years
  OS for cohort I will be analyzed as described for PFS in cohort I and OS for cohort II will be analyzed as described for PFS in cohort II. PFS of the two study arms will be compared by log-rank test (1-sided, alpha=0.1). Kaplan-Meir plot will be provided. HR and the corresponding 95% CI will be estimated by Cox proportional model using treatment as covariate. PFS for Cohort 2 will be summarized using the Kaplan-Meir's method. Median PFS with corresponding 95% CI will be provided.
Incidence of adverse events | Up to 5 years
  The grade of toxicity measurement will follow Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The distribution by treatment group of the highest grade of each CTCAEs experienced by each patient categorized will be tabulated. The tabulations will also be reviewed on a semi-annual basis by the Data Monitoring Committee. These tabulations will include summaries by system organ class and summaries by term under each system organ class.

OTHER OUTCOMES:
Analysis of integrated and exploratory biomarkers | Up to 5 years
  A separate statistical analysis plan will be developed for the integrated and exploratory biomarker analysis. Concordance of diagnostic tumor mutation profile generated by the designated laboratory, the pre-treatment biopsy mutation profile, and the pre-treatment circulating tumor deoxyribonucleic acid mutation profile will be assessed. Details are provided in the statistical plan of the ComboMATCH Registration protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Bora Lim, Principal Investigator — CenterThe University of Texas MD Anderson Cancer Center
Locations (196):
- United States (192):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Kingman Regional Medical Center, Kingman, Arizona
  - PCR Oncology, Arroyo Grande, California
  - Epic Care-Dublin, Dublin, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Saint Joseph Hospital - Orange, Orange, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Saint John Hospital - Macomb Medical, Macomb, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Memorial Hospital, Marysville, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - UPMC Altoona, Altoona, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Valley Medical Center, Renton, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
- Puerto Rico (4):
  - Puerto Rico Hematology Oncology Group, Bayamón
  - Doctors Cancer Center, Manatí
  - Centro Comprensivo de Cancer de UPR, San Juan
  - PROncology, San Juan

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT05554354/ICF_000.pdf